CLINICAL TRIAL: NCT06523712
Title: The Efficiency of an Oral Health Intervention in Promoting Better Oral Health Behaviors in Children Between the Ages of 5 to12 Years in a Low-income Nation
Brief Title: Effectiveness of Interactive Oral Care Lessons on Children Dental Health Practices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD studentship, Universiti Putra Malaysia
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UOL
Record Dates: First submitted 2024-06-15; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Intervention Model Description: In a parallel intervention study model, participants are divided into two or more distinct groups, with each group receiving a different intervention or treatment simultaneously. In this study, participants are not randomized into two arms: the experimental group (Arm 1) and the control group (Arm 2). The experimental group receives the interactive oral care lessons, while the control group does not receive any intervention and continues with their regular oral hygiene practices. Both groups are assessed at baseline and post-intervention to compare outcomes and evaluate the effectiveness of the intervention. This study design allows for the direct comparison of outcomes between the intervention and control groups, enabling researchers to determine the impact of the intervention on oral hygiene knowledge, behavior, and plaque control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this study, masking, also known as blinding, refers to the practice of concealing the allocation of participants to intervention groups from outcome assessors and investigators involved in data collection and analysis.
  Masking helps minimize bias that could occur if those assessing the outcomes are aware of the participants' assigned interventions. In this case, both the outcome assessors and investigators are masked, meaning they are unaware of which participants received the interactive oral care lessons (experimental group) and which participants were in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The participants assigned to Arm 1 will receive interactive oral care curriculum lessons designed to educate and engage them in oral hygiene practices. These lessons will cover various topics such as the importance of teeth, types of dentition, proper brushing techniques, prevention of dental caries, and the role of fluoride in maintaining oral health. The educational sessions will be delivered using interactive methods such as printed flashcards, games, and hands-on activities to enhance learning and retention. Participants will actively participate in the sessions, which will be tailored to their age group and comprehension level. The goal of Arm 1 is to assess the effectiveness of these interactive oral care lessons in improving oral hygiene knowledge, behavior, and plaque control among schoolchildren aged 5 to 12.
  Interventions: Behavioral: Smile Smarts
- Control group (No Intervention): Participants assigned to Arm 2 will serve as the control group and will not receive any intervention ( interactive oral care lessons) during the study period except basic dental hygiene education as usually practiced by schools. The purpose of Arm 2 is to serve as a comparison group to evaluate the effectiveness of the interactive oral care lessons provided to participants in Arm 1.

INTERVENTIONS:
Behavioral: Smile Smarts — The interactive oral health care lessons provided to participants in Arm 1 would involve activities and discussions aimed at changing behaviors such as tooth brushing frequency, brushing techniques, and the use of interdental aids. The intervention aims to educate and motivate participants to adopt and maintain optimal oral hygiene habits through behavioral change strategies.
  Arms: intervention group

SUMMARY:
It presents a randomized clinical trial to assess the effectiveness of interactive oral care lessons for children. It highlights the importance of oral health education during childhood and proposes using engaging teaching methods. The study involves baseline and post-intervention assessments, with participants randomly assigned to receive oral health education or serve as a control group. Data collected through questionnaires and plaque assessments will be analyzed to determine the impact of the intervention on oral hygiene habits.

DETAILED DESCRIPTION:
It presents a comprehensive research plan aimed at assessing the effectiveness of interactive oral care lessons for children through a randomized clinical trial. It begins by emphasizing the crucial role of oral health education during childhood in establishing lifelong positive oral hygiene habits. The proposed study seeks to address this need by implementing interactive teaching methods tailored to engage young learners effectively.

The study will be conducted in a schools located in Lahore.

The inclusion criteria for participant selection specify children within the age range mentioned. In contrast, exclusion criteria include those who do not provide permission and consent from both children and their parents, as well as children with underlying systemic diseases or special healthcare needs.

Data collection procedures involve obtaining approval from the departmental research committee and gaining authorization from school principals. Discussions with parents will be scheduled to explain the research in detail and obtain written consent. The schools will then be randomly divided into two groups: Group I, receiving oral health education (experimental), and Group II, serving as the control.

The study will be conducted in three phases over six months:

Phase 1: Baseline Assessment Demographic information ,oral health questionnaires will be collected. Plaque assessment will be conducted using the Silness and Loe plaque index under natural lighting conditions.

Phase 2: Intervention Group I will receive comprehensive oral health education sessions covering topics such as the importance of teeth, brushing techniques, dental caries, and preventive measures.

Group II will not receive any intervention and will serve as the control. Phase 3: Post-Intervention Assessment Oral health-related knowledge and behavior will be reassessed using the same questionnaires.

Plaque assessment will be repeated using the Silness and Loe plaque index. Data analysis will involve Intention-to-treat analysis. The Shapiro-Wilk test will be applied to explore whether the data are normally distributed. Missing data will be reported. The mean and standard deviation will be presented for normal data, whereas for non-normal data, the median and interquartile ranges will be displayed. Frequencies and percentages will be used to depict categorical data. Differences in adherence scores between the two groups at 0 and 6 months for the primary and secondary outcomes, parametric tests (Independent samples t-test/Paired samples t-test), and nonparametric tests (Mann-Whitney U test /Wilcoxon signed-rank test) will be conducted on the data. P < 0.05 will be used as the significance test. Data will be reported as to why it is missing. All analysis will be made using SPSS and R-Studio.

The outcome of the study aims to provide insights into the effectiveness of interactive oral care lessons on children dental health practices. The research schedule includes phases for data collection, data entry, data analysis, and article write-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 to 12 years. Enrollment at one of the selected schools.
* Consent obtained from parents or legal guardians for participation in the study.

Exclusion Criteria:

* Children and their parents who did not give assent and consent to participate in the study.
* Children with severe oral health issues requiring immediate medical attention.
* Children with special needs affecting their ability to participate in the oral health education interventions.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
DENTAL HEALTH PRACTICES AND BEHAVIOUR | 6 MONTHS
  The primary outcome is dental health practices and behaviour will be assessed using a pre-validated questionnaire derived from a reference study with a reliability score of 0.719. The questionnaire comprises 12 questions, where questions 1-6 pertain to awareness and questions 7-12 assess practices. The scoring range is from 0 to 12, with higher scores indicating better dental health practices and behavior.

SECONDARY OUTCOMES:
PLAQUE SCORE | 6 MONTHS
  The secondary outcome is Plaque score will be measured using the Silness and Löe plaque index. This index scores the thickness of dental plaque at the gingival margin. The scoring range is from 0 to 3, with 0 indicating no plaque and 3 indicating a high amount of plaque accumulation.
GINGIVAL SCORE | 6 MONTHS
  The other secondary outcome is gingival score will be measured using the Silness and Löe gingival index. This index assesses the severity of gingivitis based on color, consistency, and bleeding on probing. The scoring range is from 0 to 3, with 0 indicating healthy gums and 3 indicating severe inflammation.
  Scoring Criteria: Assess gingival inflammation at four sites around each tooth (mesial, distal, buccal, and lingual)
ORAL HEALTH RELATED QUALITY OF LIFE | 6 months
  Oral Health-Related Quality of Life is a vital measure that reflects the broader implications of oral health on an individual's life. By understanding and improving OHRQoL, healthcare providers and policymakers can enhance the overall health and well-being of individuals and communities.

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD ARSHED, PhD, Principal Investigator — University of Lahore

REFERENCES:
- [Result] Halawany HS, Al Badr A, Al Sadhan S, Al Balkhi M, Al-Maflehi N, Abraham NB, Jacob V, Al Sherif G. Effectiveness of oral health education intervention among female primary school children in Riyadh, Saudi Arabia. Saudi Dent J. 2018 Jul;30(3):190-196. doi: 10.1016/j.sdentj.2018.04.001. Epub 2018 May 4. PMID 29942102
- [Result] Wahengbam PP, Kshetrimayum N, Wahengbam BS, Nandkeoliar T, Lyngdoh D. Assessment of Oral Health Knowledge, Attitude and Self-Care Practice Among Adolescents - A State Wide Cross- Sectional Study in Manipur, North Eastern India. J Clin Diagn Res. 2016 Jun;10(6):ZC65-70. doi: 10.7860/JCDR/2016/20693.8002. Epub 2016 Jun 1. PMID 27504414
- [Result] Carvalho AP, Moura MF, Costa FO, Cota LO. Correlations between different plaque indexes and bleeding on probing: A concurrent validity study. J Clin Exp Dent. 2023 Jan 1;15(1):e9-e16. doi: 10.4317/jced.60039. eCollection 2023 Jan. PMID 36755682
- [Result] Hilgert LA, Leal SC, Bronkhorst EM, Frencken JE. Long-term Effect of Supervised Toothbrushing on Levels of Plaque and Gingival Bleeding Among Schoolchildren. Oral Health Prev Dent. 2017;15(6):537-542. doi: 10.3290/j.ohpd.a39593. PMID 29319063
- [Result] Pine C, Adair P, Robinson L, Burnside G, Moynihan P, Wade W, Kistler J, Curnow M, Henderson M. The BBaRTS Healthy Teeth Behaviour Change Programme for preventing dental caries in primary school children: study protocol for a cluster randomised controlled trial. Trials. 2016 Feb 20;17(1):103. doi: 10.1186/s13063-016-1226-3. PMID 26897029
- [Result] Florio FM, Dos Santos Klee L, Brandao Ramos AP, Ambrosano GMB, de Souza Fonseca Silva A. Use of Water by Schoolchildren: Impact of Indirectly Supervised Daily Toothbrushing-A Pilot Study. Int J Clin Pediatr Dent. 2020 Sep-Oct;13(5):513-517. doi: 10.5005/jp-journals-10005-1800. PMID 33623340
- [Result] Salama FS, Al-Balkhi BK. Effectiveness of educational intervention of oral health for special needs on knowledge of dental students in Saudi Arabia. Disabil Health J. 2020 Jan;13(1):100789. doi: 10.1016/j.dhjo.2019.03.005. Epub 2019 Mar 19. PMID 31495647
- [Result] Swe KK, Soe AK, Aung SH, Soe HZ. Effectiveness of oral health education on 8- to 10-year-old school children in rural areas of the Magway Region, Myanmar. BMC Oral Health. 2021 Jan 2;21(1):2. doi: 10.1186/s12903-020-01368-0. PMID 33388030
- Available data/document: Informed Consent Form — https://schoolsplus.pk/schools/sharif-education-complex/
- Available data/document: Informed Consent Form — https://apseducation123.wixsite.com/website
- Available data/document: Informed Consent Form — https://apsaskarixi.pk/